CLINICAL TRIAL: NCT02379884
Title: Mechanical Ventilation in Internal Medicine Elderly Patients - Choosing Wisely
Acronym: VentWise
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Israel National Institute for Health Policy and Health Services Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0399-14-RMB CTIL
Record Dates: First submitted 2015-02-22; First posted 2015-03-05 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Arrest
Keywords: Mechanical ventilation; Elderly; Mortality; Health services
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective observational study evaluating all patients requiring mechanical ventilation. Data will be gathered regarding the events prior to ventilation and the indication for mechanical ventilation. In-hospital and post-admission outcome will be monitored.

DETAILED DESCRIPTION:
Background The aging of the population associated with increased morbidity, on one hand, and technological advances providing life-sustaining treatments on the other, resulted in an increased number of mechanically ventilated patients in Internal Medicine wards. In a previous study the investigators found that about half of the hospitalization days in intermediate care units in Internal Medicine wards were utilized by older patients at the end of life. The mortality at 6 months from the time of admission was greater than 70%, unrelated to the type of treatment. The majority of the elderly patients surviving the acute stage were transferred to chronic long-term care hospitals. The Public Health System in Israel invests costly resources in providing care to mechanically ventilated patients in both acute and chronic care settings, in spite of unproved benefit on the quality of life and on life expectancy.

Aims of the study

1. Identification of patients and the factors affecting the decision-making process and outcome in mechanically ventilated patients in Internal Medicine wards in acute care hospitals.
2. Development of a predictive model to classifying mechanically ventilated patients by outcome on the basis of patient characteristics on admission and the factors involved in decision-making.
3. Assessment of medical resource investment according to the study model groups.

Study hypothesis Identification of parameters predicting better outcome and potential for rehabilitation in elderly mechanically ventilated internal medicine patients, versus patients with poorer outcome who would need palliative care.

Methods The study is a prospective observational study carried out in five Internal Medicine wards and the Medical Intensive Care Unit at the Rambam Health Care Campus in Haifa, Israel. All patients requiring mechanical ventilation will be included. Patients' medical and demographic data will be obtained from the hospital computerized record system. Data will be gathered regarding the events prior to ventilation and the indication for mechanical ventilation. In-hospital and post-admission outcome will be monitored. Mortality at 6 months will be obtained from the Israel National Population Registry. Descriptive statistical analysis will be performed, and multivariate logistic regression analysis will be applied to identify variables contributing to the need for ventilation and outcome.

Importance of the study The approval of the 2005 Dying Patient Act in Israel, allowed for withholding of certain life-sustaining interventions at end of life. However, once an intervention such as mechanical ventilation has been commenced, the Law does not permit its withdrawing, making the decision to ventilate a patient irreversible. There is thus a clear need to improve the decision-making process related to undertaking mechanical ventilation in elderly internal medicine patients. In addition, the investigators believe that the study will highlight the issue and bring the policy makers to the establishing practical tools for health care professionals. The investigators also hope that the study will incite the general public attention to address the issue of advanced directives regarding undergoing invasive treatments such as mechanical ventilation at end of life. Finally, the investigators consider that adoption of a more evidence-based approach to undertaking mechanical ventilation, and consideration of patients' advanced directives, by health care providers in both community and in-patient settings, will lead to a better utilization of health resources and improvement of end of life of care.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation
* Males and females
* Age over 18 years
* Admitted to internal medicine wards or medical intensive care unit

Exclusion Criteria:

* Younger than 18 years
* Surgical and trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients requiring mechanical ventilation over the study period.
  Inclusion criteria:
  Males and females Age over 18 years Admitted to internal medicine wards or medical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of randomization until the date of first documented date of death from any cause, assessed up to 6 months
  Data will be obtained from the Israel National Population Registry

SECONDARY OUTCOMES:
Length of acute hospital stay | From date of randomization until the date of first documented discharge from the acute care hospital to the community or to a long-term care institution, assessed up to 6 months
  Data will be obtained from the acute care hospital computerized record system
Ongoing medical and nursing care in a long term care institution | From date of randomization until the date of first documented discharge from the acute care hospital to a long-term care institution, assessed up to 6 months
  Data will be obtained from the acute care hospital computerized record system

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD MBBCh, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No